CLINICAL TRIAL: NCT04092465
Title: Short and Long Term Outcomes of Patients With Locally Advanced Non-Small Cell Lung Cancer Undergoing Pulmonary Parenchyma Resection After Induction Treatment.
Brief Title: Outcomes of Surgical Resection After Induction Treatment in Non-Small Cell Lung Cancer (SRaIT)
Acronym: SRaIT
Status: Completed | Type: Observational
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Christophoros N. Foroulis, Associate Professor of Thoracic Surgery, AHEPA University Hospital
Other Study IDs: 425/12-9-2019
Record Dates: First submitted 2019-08-31; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Patient Outcome Assessment; Morbidity; Mortality
Keywords: NSCLC; Locally Advanced NSCLC; Induction treatment; Induction chemotherapy; Induction chemoradiotherapy; Pulmonary Parenchyma Resection; Surgical Outcomes; Survival; Morbidity; Thoracotomy
MeSH Terms: interventions — Pneumonectomy; Induction Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pulmonary parenchyma resection, lobectomy, pneumonectomy, sleeve lobectomy, extended lobectomy/pneumonectomy — Resection of the downstaged locally advanced NSCLC through formal thoracotomy
  Other Names: induction chemotherapy, induction chemoradiotherapy

SUMMARY:
Surgery still remains the main treatment option for Non-Small Cell Lung Cancer (NSCLC) which is limited within the lung parenchyma and possibly invades the intrapulmonary or hilar nodes. The role of surgery in locally advanced NSCLC with the form of invasion of adjacent strictures or mediastinal nodes is a 30-year point of discussion and debate among thoracic surgeons, clinical and radiation oncologists, chest physicians and other related specialties. Despite the continuous debate the management of locally advanced NSCLC varies between different countries and different institutions.We try to investigate the short and long term outcomes of surgery after induction treatment performed for locally advanced NSCLC.

DETAILED DESCRIPTION:
All patients who underwent surgery with curative intent or salvage after induction treatment during a 8-year time period (2011-2019). Induction treatment with the form either of chemotherapy or chemoradiotherapy was delivered according to the thoracic multidisciplinary team decision which it was based on primary tumor histology and stage. Patients with Pancoast tumors were excluded from the study design, because these tumors have different clinical characteristics and represent a separate category of NSCLC with a well recognized specific treatment plan worldwide.

Overall 42 patients are included in the study and the recorded parameters in each patient are:

1. Age, gender, comorbidities, histology, location in the lung and stage of tumor at presentation, tools used for preoperative staging in each case, any previous surgical procedures of other treatments performed before elsewhere, type of induction treatment, tools used for tumor restaging.
2. In each patient were recorded any specific technical details concerning the applied surgical procedures, time of surgery and one-lung ventilation (OLV), postoperative complications and their management, mortality, pos-resection staging (ypTNM), the number of resected lymph nodes in each patient.
3. Concerning the long term outcomes, overall and disease-free survival, kind of recurrence (local, distant, combination) and treatment of recurrences were recorded.

Interpretation fo the results will include the correlation of surgical details, kind and dose of induction treatment with postoperative complications, especially infectious complications and prolonged air leaks. Radicality of the resection and response of the tumor to induction treatment (ypTNM stage) as it is recorded in histology reports are the two important clinical parameters to be studied for their effect on long term survival and recurrences.

Surgery was applied as salvage surgery in not well responded tumors or as resection of downstaged tumors.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent surgery for NSCLC after induction treatment

Exclusion Criteria:

Patients who underwent surgery fo NSCLC located in the superior sulcus and Pancoast syndrome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent resection with curative intent of their locally advanced NSCLC after induction treatment in a single Academic Center from September 2011 to August 2019 (8 years). Surgery was applied either in downstaged tumors os as salvage extended surgery in patients not responding to induction treatment.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2011-09-30 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Mortality-Morbidity | From date of surgery until 12 weeks after surgery
  Mortality and morbidity of the pulmonary parenchyma resection for NSCLC after induction treatment
Long term survival of patients and correlation of long term survival with the post-resection stage of tumor (ypTNM stage) | From the date of surgery to up to 96 months after surgery
  Close clinical follow-up by clinical oncologists and surgeons to detect and treat
Recurrence of tumor - Disease free survival | From date of surgery to up to 96 months after surgery
  Close clinical follow-up by clinical oncologists and surgeons to detect and treat recurrences. Correlation of recurrences with post-resection (ypTNM) stage of tumor, completeness of resection, type of surgical procedure

SECONDARY OUTCOMES:
Specific details concerning the surgical procedures and correlation with morbidity | From time of surgery to up to 12 weeks after surgery
  Extended procedures, intrapericardial procedures, pneumonectomy
Respiratory complications | From time of surgery to up to 12 weeks after surgery
  Correlation of the overall time required for the procedure and of the time of one lung ventilation with the rate and kind of respiratory complications and ICU stay
Postoperative complications | From time of surgery to up to 12 weeks after surgery
  Correlation of kind and overall dose of the delivered chemotherapy or radiotherapy with the development of postoperative complications, especially prolonged air leak and infectious complications

CONTACTS AND LOCATIONS:
Overall Officials: CHRISTOFOROS N FOROULIS, Professor, Principal Investigator — AHEPA University Hospital; KYRIAKOS ANASTASIADIS, Professor, Principal Investigator — AHEPA University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shepherd FA. Induction chemotherapy for locally advanced non-small cell lung cancer. Ann Thorac Surg. 1993 Jun;55(6):1585-92. doi: 10.1016/0003-4975(93)91123-5. PMID 8390231
- [Background] Rusch VW, Albain KS, Crowley JJ, Rice TW, Lonchyna V, McKenna R Jr, Livingston RB, Griffin BR, Benfield JR. Surgical resection of stage IIIA and stage IIIB non-small-cell lung cancer after concurrent induction chemoradiotherapy. A Southwest Oncology Group trial. J Thorac Cardiovasc Surg. 1993 Jan;105(1):97-104; discussion 104-6. PMID 8380477
- [Background] Albain KS, Rusch VW, Crowley JJ, Rice TW, Turrisi AT 3rd, Weick JK, Lonchyna VA, Presant CA, McKenna RJ, Gandara DR, et al. Concurrent cisplatin/etoposide plus chest radiotherapy followed by surgery for stages IIIA (N2) and IIIB non-small-cell lung cancer: mature results of Southwest Oncology Group phase II study 8805. J Clin Oncol. 1995 Aug;13(8):1880-92. doi: 10.1200/JCO.1995.13.8.1880. PMID 7636530
- [Background] Sonett JR, Suntharalingam M, Edelman MJ, Patel AB, Gamliel Z, Doyle A, Hausner P, Krasna M. Pulmonary resection after curative intent radiotherapy (>59 Gy) and concurrent chemotherapy in non-small-cell lung cancer. Ann Thorac Surg. 2004 Oct;78(4):1200-5; discussion 1206. doi: 10.1016/j.athoracsur.2004.04.085. PMID 15464470
- [Background] Kumar P, Herndon J 2nd, Langer M, Kohman LJ, Elias AD, Kass FC, Eaton WL, Seagren SL, Green MR, Sugarbaker DJ. Patterns of disease failure after trimodality therapy of nonsmall cell lung carcinoma pathologic stage IIIA (N2). Analysis of Cancer and Leukemia Group B Protocol 8935. Cancer. 1996 Jun 1;77(11):2393-9. doi: 10.1002/(SICI)1097-0142(19960601)77:113.0.CO;2-Q. PMID 8635112